CLINICAL TRIAL: NCT02509793
Title: A Pilot Study Assessing Impulsivity in Patients With Huntington's Disease on Xenazine (Tetrabenazine)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: William Ondo, MD (Other)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor-Investigator, William Ondo, MD, Professor, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013929; HSC-MS-13-0878 (Other: UTHealth -Houston)
Record Dates: First submitted 2015-07-24; First posted 2015-07-28 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — Tetrabenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tetrabenazine (Experimental): Xenazine (tetrabenazine), pill, dosage titrated to effect, three times a day, 12 weeks
  Interventions: Drug: Tetrabenazine

INTERVENTIONS:
Drug: Tetrabenazine — Xenazine, pill, dose to effect, three times a day, for 12 weeks
  Other Names: Xenazine

SUMMARY:
The purpose of this research study is to see if tetrabenazine, which is commonly used to treat Huntington's Disease (HD), reduces the problems of impulsivity that are common in patients with HD. Investigators will also see how the medicine affects aspects of thinking and mood.

DETAILED DESCRIPTION:
This study is an open-label assessment of behavioral symptoms including depression, impulsivity, and suicidal ideations in patients prior to, and after, taking a stable dose of TBZ for Huntington's disease. All subjects will be evaluated with tests of depression (Beck Depression Scale), impulsivity (QUIP, BIS-11, and computerized impulsivity scales), and suicidal ideation (Columbia Suicide Scale) as a safety measure before they actually start taking TBZ. Since there is a significant lack of awareness of emotional and cognitive symptoms (anosagnosia) in patients with HD, collateral sources will be asked to fill out similar questionnaires based on their knowledge and observation of the patient. Patients and collaterals will be asked to return to the clinic for an identical evaluation plus adverse events, after they have been on a stable dose of TBZ for 4 weeks, which would be 8 ± 1 week after initiating TBZ. Patients will be titrated over 3-5 weeks to best dose as determined by the investigator, up to a maximum of 75 mg/day. As patients are titrating, there will be several telephone contacts conducted. The initial dose will be 12.5 mg BID. Best dose will be largely determined by adverse events and subjective efficacy. Determination of best dose will include two scheduled phone calls and others as needed. Other medications will remain stable between visits.

ELIGIBILITY:
Inclusion Criteria:

* For HUntington's Disease (HD) patients only--Definite HD as indicated by positive gene testing or typical symptoms in the context of family history of HD.
* A moderate degree of impulsivity as measured by the Barrat Impulsivity Scale (BIS). (>65)
* Must be symptomatic in the opinion of the investigator. Standard clinical criteria for symptomatic HD will be employed, any motor signs c/w HD, usually chorea.
* Patient is cognitively alert and able to answer/understand.

Exclusion Criteria:

* Patient requires the assistance of another person to walk, or is non-ambulatory.
* Patient is severely impaired cognitively.
* Patients taking neuroleptic (dopamine blocking) medications within the past 14 days.
* patient is actively suicidal, has untreated or inadequately treated depression, has impaired hepatic function, is taking MAO inhibitors or is taking reserpine or has been off of reserpine for less than 20 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Score on the Questionnaire for Impulsive Disorders in Parkinson's Disease | Baseline and 8 weeks
  A newly developed and tested tool for measuring impulsivity in PD patients.
Change in Score on the Geriatric Depression Scale | Baseline and 8 weeks
  This assessment detects depressive symptoms in subjects and is a commonly used neuropsychological scale. It is less influenced by motor / somatic symptoms compared to other depression scales.
Change in Score on the Barrat Impulsivity Scale | Baseline and 8 weeks
  Scale is the most widely used self-report measure of impulsive personality traits. The BIS-11 is a 30-item self-report questionnaire that is scored to yield a total score, three second-order factors, and six first-order factors.
Change in Score on the Minnesota Impulsivity Disorders Interview | Baseline and 8 weeks
  This is a clinician-administered screening instrument that had shown good reliability and validity in studies of adult and adolescent psychiatric patients.
Change in Score on the Iowa Gambling Task | Baseline and 8 weeks
  a widely used, but complex, neuropsychological task of executive function in which mixed outcomes (gains and losses) are experienced together, to performance on a relatively simpler descriptive task, the Cups task, which isolates adaptive decision making for achieving gains and avoiding losses. It is very predictive of impulsive personality traits
Change in Score on the Montreal Cognitive Impairment Assessment | Baseline and 8 weeks
  cognitive screening test designed to assist Health Professionals for detection of mild cognitive impairment, including Alzheimer's disease.

SECONDARY OUTCOMES:
Change in Score on the United Huntington's Disease Rating Scale - Motor section | Baseline and 8 weeks
  A clinical examination of various cognitive, behavioral, and motor features commonly seen in patients with HD (Huntington Study Group, 1996). This is a standardized test used in most clinical studies of HD.

CONTACTS AND LOCATIONS:
Overall Officials: William G Ondo, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Neurological Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided